CLINICAL TRIAL: NCT06292364
Title: "Comparison of Retention Characteristics of Immediate vs Delayed Retainer Delivery Using 3 Dimensional Digital Model Analysis : A Prospective Clinical Trial "
Brief Title: Comparison of Retention Characteristics of Immediate vs Delayed Retainer Delivery Using 3D Digital Model Analysis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PGIDS/BHRC/23/106
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Relapse
Keywords: orthodontic retention
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): beggs wrap around Retainer will be given to the patients immediately [Just after debonding].
  Interventions: Other: immediate orthodontic retainer delivery
- experimental group (Active Comparator): beggs wrap around Retainer will be delivered to the patients 7 days post debonding.
  Interventions: Other: delayed orthodontic retainer delivery

INTERVENTIONS:
Other: immediate orthodontic retainer delivery — post orthodontic treatment patients will be given orthodontic retainer immediately after debonding
  Arms: control group
Other: delayed orthodontic retainer delivery — post orthodontic treatment patients will be given orthodontic retainer after 7 days of debonding
  Arms: experimental group

SUMMARY:
Retention has been defined as "the holding of teeth following orthodontic treatment in the treated position for the period of time necessary for the maintenance of the result". Controversies regarding retention regime exist due to lack of high quality evidence regarding duration, type and timing of different type retainer.The present randomised controlled trial will be undertaken to assess the changes and compare if there is any difference in movement of teeth in post orthodontic treatment cases with immediate and delayed (post 7 days) delivery using beggs retainer and change in level of bone biomarker over 6 months period of retention .

DETAILED DESCRIPTION:
The proposed study will be a prospective, non-pharmacological, single blind, randomized clinical trial to evaluate if there is a difference in transverse (X-axis), A-P(Y-axis) and Vertical plane(Z-axis) of dentition in two group of post orthodontic treatment patients with immediate retainer delivery(Beggs wrap around retainer ) in one group and post 7 days retainer delivery( beggs wrap around retainer) in other group of patients. The present study will be conducted in the Department of Orthodontic and Dentofacial Orthopedics, P.G.I.D.S, Pt. B.D Sharma University of health sciences, Rohtak. The study will be carried out after the institutional approval obtained from ethical committee.

A sample size of 18 patients was calculated keeping confidence interval 95% with power 80%. Accounting for a 10% drop out rate, 20 patients will be enrolled in each group. Patient will be randomly allocated to the study group by a person not involved in the trial using computer generated randomization list. Changes in the tooth movement in transverse(X-axis), A-P(Y-axis), Vertical plane(Z-axis) will be compared in terms of intercanine width, intermolar width, overjet, overbite and contact point displacement between the two groups at following time intervals. These parameters will be charted at T0, T1, T2,T3 and T4 for each patient.Changes in the tooth movement in transverse(X-axis), A-P(Y-axis), Vertical plane(Z-axis) will be compared in terms of intercanine width, intermolar width, overjet, overbite and contact point displacement between the two groups at following time intervals. These parameters will be charted at T0, T1, T2,T3 and T4 for each patient. T0 - Baseline records, at the time of debonding. T1 - Records obtained at the time of retainer delivery. T2 - Records obtained after 1 month of retainer delivery. T3 - Records obtained after 3 months of retainer delivery. T4 - Records obtained after 6 months of retainer delivery

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who required extraction.
2. Optimal functional occlusion at end of treatment (PAR score >70%).
3. Littles irregularity index (Pre-treatment <6mm in both upper and lower arch).
4. Nonsurgical and non-orthopedic patients.
5. Non syndromic patients and no impaction of teeth except third molars.
6. Optimal periodontal condition and Good oral hygiene (probing depth <3mm, gingival index score <1
7. Good compliance regarding retainer wear.

Exclusion Criteria:

1. Subjects with incomplete orthodontic treatment.
2. TMJ disorder patients.
3. Any systemic disease affecting bone and general growth.
4. Patients with incomplete records.
5. Patient who fail to follow up or undergo complete treatment.
6. Patient with learning difficulties
7. Patients having antibiotic therapy within previous 3 months and used anti inflammatory drugs in the month before the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-05 (Actual); Primary Completion 2024-11-05 (Estimated); Study Completion 2024-12-05 (Estimated)

PRIMARY OUTCOMES:
overjet | T0 - baseline on the day of debonding
  sagittal distance between upper and lower incisors
overjet | T1 - 7 days after debonding
  sagittal distance between upper and lower incisors
overjet | T2 - 1 month after debonding
  sagittal distance between upper and lower incisors
Overjet | T3 - 6 month after debonding
  sagittal distance between upper and lower incisors
contact point displacement | T0 - baseline on the day of debonding
  displacement of contact points in anterior teeth
contact point displacement | T1 - 7 days after debonding
  displacement of contact points in anterior teeth
contact point displacement | T2 - 1 month after debonding
  displacement of contact points in anterior teeth
contact point displacement | T3 - 6 month after debonding
  displacement of contact points in anterior teeth
overbite | T0 - baseline on the day of debonding
  vertical overlap of upper and lower incisors
overbite | T1 - 7 days after debonding
  vertical overlap of upper and lower incisors
overbite | T2 - 1 month after debonding
  vertical overlap of upper and lower incisors
overbite | T3 - 6 month after debonding
  vertical overlap of upper and lower incisors
intermolar width | T0 - baseline on the day of debonding
  transverse distance between the first molars
intermolar width | T1 - 7 days after debonding
  transverse distance between the first molars
intermolar width | T2 - 1 month after debonding
  transverse distance between the first molars
intermolar width | T3 - 6 month after debonding
  transverse distance between the first molars
intercanine width | T0 - baseline on the day of debonding
  transverse distance between the canine
intercanine width | T1 - 7 days after debonding
  transverse distance between the canine
intercanine width | T2 - 1 month after debonding
  transverse distance between the canine
intercanine width | T3 - 6 month after debonding
  transverse distance between the canine

SECONDARY OUTCOMES:
GCF - elisa | Tb - 1 month before debonding
  BALP AND CTX TYPE 1 BIOMARKER
GCF - elisa | T0 - on the day of debonding
  BALP AND CTX TYPE 1 BIOMARKER
GCF - elisa | T1 - 1 week after debonding
  BALP AND CTX TYPE 1 BIOMARKER
GCF - elisa | T2 - 1 month after debonding
  BALP AND CTX TYPE 1 BIOMARKER

CONTACTS AND LOCATIONS:
Locations (1):
- Pgids Rohtak, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No